CLINICAL TRIAL: NCT04248231
Title: The CINSARC Genomic Signature as a Predictor of Resectability of High Grade Serous Ovarian Adenocarcinomas
Brief Title: CINSARC Genomic Signature as Predictor of Resectability of Ovarian Adenocarcinoma
Acronym: OVASARC
Status: Completed | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 18HLGENF05
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CINSARC signature — CINSARC molecular signature analysis

SUMMARY:
The majority of primary cancers of the ovary or peritoneum are represented by high-grade serous adenocarcinomas. These are rare pathologies, the incidence of which is estimated at 7.1 per 100,000, representing approximately 4,500 new cases per year in France (INCA 2017). In the absence of effective screening, nearly 85% of patients have an advanced disease at diagnosis (corresponding to the FIGO III or IVA stage, characterized by diffuse peritoneal involvement). Despite multidisciplinary care, the majority of patients (80%) will recur within a median of 18 to 24 months.

It is therefore necessary to develop new tools, in particular molecular, in order to allow :

* to better select patients accessible to full interval surgery
* to exclude patients who would not benefit from this surgery in terms of survival

In 2010, Chibon et al. identified, from a cohort of patients with soft tissue sarcoma (STM), a molecular signature (called CINSARC), based on the expression profile of 67 genes involved in mitotic control and chromosomal integrity. The team showed that this transcriptomic signature is an independent prognostic factor in different types of STM, but also a prognostic factor more discriminating than the histological grade (FNCLCC), historical and major prognostic factor of STM.

Being initially made from frozen material and on a DNA biochip (Affymetrix), this signature was unusable outside the field of fundamental research. This is why CINSARC has been gradually optimized, first by the RNA sequencing technique on frozen tissue fixed in formalin (FFPE), and recently on FFPE tissue by the NanoString® technique. This very sensitive and inexpensive technique requires only small amounts of total RNA, making it compatible with use on "routine" diagnostic samples, microbiopsy or surgical biopsy, opening the door to real clinical application. Several clinical studies using this latest CINSARC optimization (called NanoCind®) to determine the treatment of patients with STM will also begin soon.

As a result of this work, necessary in order to more precisely support the potential of CINSARC in this pathology, the investigators hope to be able to assess from the diagnosis the evolutionary potential of the patients, which could make it possible to evaluate therapeutic strategies adapted to the profiles of each subpopulation: the investigators can for example imagine in theory a therapeutic de-escalation for low-risk patients, or else, for very high-risk patients, an intensified strategy.

DETAILED DESCRIPTION:
RNA extraction from 150 patients archival tumor, fragments of 50 to 300 nucleotides size.

RNA preparation, hybridation, detection, scanning according to Nanostring manufacturer recommandations: obtention of CINSARC molecular signature Sensibility, specificity, prognostic value of the signature will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian adenocarcinoma treated in IUCTO Toulouse by primary chemotherapy and for whom diagnosis tumoral sample is available

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study on medical, clinical, pathologic data from patients primary treated for ovarian adenocarcinoma . 150 cases analyzed
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
The main endpoint is the sensitivity of the CINSARC signature to identify surgical resectability after neoadjuvant chemotherapy. | sept 2019-sept 2020
  Sensitivity (Se), is defined by the proportion of subjects defined as Low risk by the CINSARC signature and having been resected, among the subjects having been resected

SECONDARY OUTCOMES:
Specificity of the CINSARC signature | sept 2019-sept 2020
  Proportion of subjects defined as high risk by the signature and having not been resected among patients having not been resected
Positive predictive value of the signature | sept 2019-sept 2020
  Proportion of subjects defined as Low risk by the signature among all subjects
Negative predictive value of the signature | sept 2019-sept 2020
  Proportion of subjects defined as High risk by the signature among all subjects
Global survival | sept 2019-sept 2020
  Time frame between diagnosis date of advanced stage / metastatic stage and date of death or last news
Progression Free survival | sept 2019-sept 2020
  Time frame between date of diagnosis of advanced stage / metastatic stage and date of either progression or death or last news

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius Regaud Institut Universitaire du cancer Toulouse Oncopole, Toulouse, France